CLINICAL TRIAL: NCT05996484
Title: Anlotinib in Combination With Toripalimab and Chemotherapy for Neoadjuvant Treatment of Resectable Esophageal Squamous Cell Carcinoma: a Phase II Clinical Study
Brief Title: Neoadjuvant Therapy of Anlotinib Combined With Toripalimab and Chemotherapy for Resectable Esophageal Carcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NFEC-2023-310
Record Dates: First submitted 2023-08-10; First posted 2023-08-18 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Esophageal Carcinoma; Neoadjuvant Therapy
MeSH Terms: conditions — Esophageal Neoplasms | interventions — toripalimab; anlotinib; Paclitaxel; Injections; Cisplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neoadjuvant Anlotinib Combined With Toripalimab and Chemotherapy (Experimental): Toripalimab+ Anlotinib+Albumin-bound paclitaxel+Cisplatin
  Interventions: Drug: Toripalimab; Drug: Anlotinib hydrochloride; Drug: Albumin paclitaxel; Drug: Cisplatin

INTERVENTIONS:
Drug: Toripalimab — Toripalimab, 240mg, IV., D1, every 3 weeks, 4 cycles.
  Other Names: JS001
Drug: Anlotinib hydrochloride — Anlotinib Hydrochloride is a capsule in the form of 8 mg ,10 mg and 12 mg, orally, once daily, 2 weeks on/1 week off, every 3 weeks, 4 cycles.
  Other Names: Anlotinib
Drug: Albumin paclitaxel — Albumin paclitaxel, 200-260 mg/m2, IV., D1, every 3 weeks, 4 cycles.
  Other Names: Paclitaxel For Injection (Albumin Bound)
Drug: Cisplatin — Cisplatin, 60-75 mg/m2, IV., D1, every 3 weeks, 4 cycles.
  Other Names: CDDP

SUMMARY:
The purpose of this study is to explore the effectiveness and safety of the combination of Anlotinib, Toripalimab, and albumin-bound paclitaxel with cisplatin for neoadjuvant therapy in resectable esophageal squamous cell carcinoma. The study aims to improve the pathological complete response rate (pCR), R0 resection rate, and disease-free survival (DFS) in patients undergoing esophageal cancer surgery. The findings of this study will provide guidance and new options for the treatment of locally advanced esophageal cancer patients.

DETAILED DESCRIPTION:
Both anti-angiogenic therapy and immune checkpoint inhibitors have shown preliminary efficacy and safety data in the field of neoadjuvant therapy for esophageal cancer. However, there is currently no available data on the combination of immune checkpoint inhibitors, anti-angiogenic therapy, and chemotherapy in neoadjuvant therapy for esophageal cancer. Based on the favorable survival benefits of this combination in first-line and second-line treatments for multiple tumors, we aim to explore another neoadjuvant treatment approach - adding anti-angiogenic agents to immune checkpoint inhibitor-based neoadjuvant therapy, providing a new perioperative treatment strategy for esophageal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age range: 18-70 years, both male and female.
2. Patients with histopathological diagnosis of esophageal squamous cell carcinoma confirmed by gastroscopy/ultrasound gastroscopy, and clinical diagnosis of cT2N1-2M0 or cT3N0-2M0, with TNM staging of stage II-III B.
3. Non-cervical esophageal cancer patients.
4. No prior systemic or local treatment for esophageal cancer, with at least one measurable lesion for imaging evaluation of neoadjuvant therapy according to RECIST 1.1 criteria.
5. ECOG PS (Eastern Cooperative Oncology Group Performance Status): 0-1.
6. Estimated survival period ≥12 months.
7. Subjects without significant dysfunction of major organs, with normal assessment of thyroid, lung, liver, kidney, and cardiac function.
8. Reproductive-age women must have taken reliable contraceptive measures or undergone pregnancy testing (serum or urine) within 7 days prior to enrollment, with negative results, and be willing to use appropriate contraception during the trial and for 8 weeks after the last administration of the investigational drug. For males, they must agree to use appropriate contraception during the trial and for 8 weeks after the last administration of the investigational drug, or have undergone surgical sterilization.
9. Subjects voluntarily participate in this study, sign an informed consent form, demonstrate good compliance, adhere to the planned schedule for regular clinical follow-up and necessary treatment, and cooperate in obtaining regular blood and tissue samples.

Exclusion Criteria:

1. Patients who have had or currently have other malignant tumors within the past 1.5 years, except for cured cervical carcinoma in situ, non-melanoma skin cancer, and superficial bladder tumors [Ta (non-invasive tumor), Tis (carcinoma in situ), and T1 (tumor invades lamina propria)].
2. Patients with ulcerative esophageal squamous cell carcinoma.
3. Patients with esophageal fistula or tracheal fistula.
4. Patients allergic to anlotinib, toripalimab, or albumin-bound paclitaxel.
5. Patients with a history of immunodeficiency diseases, including HIV-positive patients or those with other acquired or congenital immunodeficiency diseases, or a history of organ transplantation.
6. Patients with severe and/or uncontrolled diseases are excluded from the study, including:

   6.1 Patients with unsatisfactory blood pressure control (systolic blood pressure ≥160 mm Hg or diastolic blood pressure ≥100 mmHg).

   6.2 Patients with grade I or higher myocardial ischemia or myocardial infarction.

   6.3 Patients with arrhythmia (including QT interval ≥480 ms) and grade I heart failure.

   6.4 Patients with poorly controlled diabetes (fasting blood glucose >10 mmol/L) or receiving high-dose glucocorticoid therapy.

   6.5 Patients with active or uncontrolled severe infections. 6.6 Patients with decompensated liver disease, active hepatitis B (HBV-DNA ≥10^4 copies/ml or 2000 IU/ml), or hepatitis C (positive for hepatitis C antibodies and HCV RNA) exceeding the lower limit of the analytical method.

   6.7 Patients with hyperthyroidism or hypothyroidism. 6.8 Patients with active tuberculosis.
7. Unresolved toxicities of grade 2 or higher, excluding alopecia, caused by any prior treatment.
8. Individuals with multiple factors that affect oral medication administration, such as dysphagia, chronic diarrhea, and intestinal obstruction.
9. Individuals with urine routine showing urinary protein ≥++, and confirmed 24-hour urine protein quantification >1.0 g.
10. Individuals who underwent major surgical treatment, incisional biopsy, or significant traumatic injury within 28 days prior to randomization.
11. Abnormal coagulation function: INR >1.5 or prothrombin time (PT) > ULN + 4 seconds or APTT > 1.5 ULN, with a bleeding tendency or receiving thrombolytic or anticoagulation therapy. Patients who experienced any bleeding or hemorrhagic events ≥ grade 3 CTCAE within 4 weeks prior to randomization, with unhealed wounds, ulcers, or fractures.
12. Occurrence of arterial/venous thrombotic events within 6 months, such as cerebrovascular accidents (including transient ischemic attacks), deep vein thrombosis, and pulmonary embolism.
13. Pregnant or lactating women.
14. Presence of distant metastasis.
15. Patients with significant bone marrow suppression.
16. Patients with mental illness or a history of substance abuse with psychotropic drugs.
17. Patients who participated in other drug clinical trials within 4 weeks.
18. Patients with accompanying diseases that, in the investigator's judgment, pose a serious risk to patient safety or may affect the patient's completion of the study.
19. Patients with inherited bleeding tendencies, coagulation disorders, potential invasion of major blood vessels, and other bleeding risks, who experienced clinically significant bleeding symptoms or had a clear bleeding tendency with gastrointestinal bleeding, bleeding gastric ulcers, baseline fecal occult blood ++ and above within 3 months prior to enrollment.
20. Patients deemed unsuitable

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Pathologic complete remission (PCR) | Immediately after the surgery
  Primary tumor or lymph node surgery specimen pathological examination without residual tumor cell

SECONDARY OUTCOMES:
R0 resection rate | Immediately after the surgery
  Residual tumor rate
Objective response rate (ORR) | Up to 36 month
  ORR is defined as the percentage of participants in the analysis population who have a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: ≥30% decrease in the sum of diameters of target lesions) per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1
Disease control rate (DCR) | Up to 36 month
  DCR is defined as the percentage of participants in the analysis population who have a CR, PR or stable disease (SD) per RECIST 1.1.
Disease-free survival (DFS) | 3(5) years after last patient enrolled
  Survival without local or systemic recurrence
Overall survival (OS) | Up to 36 month
  Overall survival is defined as the duration from date of enrollment to the date of death from any cause.
Safety: AE | Up to 36 month
  Safety was defined as the Number of Participants With an Adverse Event
Change From Baseline in HRQoL Score Using EORTC Quality of Life Questionnaire-Oesophageal Module (QLQ-OES18) | Up to 36 month
  The EORTC QLQ-OES18 is a disease-specific questionnaire to assess measurements specific to esophageal cancer. It contains 18 items and is based on four subscales-dysphagia, eating, reflux and pain. All items are scored using a four-point scale that offers these response choices: 1=not at all, 2=a little, 3=quite a bit, 4=very much. A higher score indicates worse level of symptoms. Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. The change from baseline in HRQoL QLQ-OES18 score in participants will be presented.

CONTACTS AND LOCATIONS:
Overall Officials: kaican cai, M.D., PhD, Principal Investigator — Nanfang Hospital, Southern Medical University

IPD SHARING:
Plan to Share IPD: No